CLINICAL TRIAL: NCT02799225
Title: Prevalence of Clinical Strains of Enterobacteria With Reduced Susceptibility to Carbapenems in the North-West Region of France
Acronym: ERC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PHRCIR11-DR-MAMMERI
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Enterobacteriaceae
Keywords: carbapenems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Enterobacteria

SUMMARY:
Enterobacteria constitute a family of Gram negative bacilli of the gastrointestinal flora. These micro-organisms are frequently responsible for nosocomial or community-acquired infections, for which treatment is essentially based on the use of beta-lactam antibiotics. This class of antibiotics comprises penicillins, cephalosporins, monobactams and carbapenems. Carbapenems have the advantage of possessing a broad antibacterial spectrum and the capacity to resist the hydrolytic action of a large number of beta-lactamases, widespread inactivating enzymes.

However, new enzymes, called carbapenemases, able to confer resistance to carbapenems either alone or in combination with additional resistance mechanisms such as loss of membrane permeability or overexpression of efflux systems, are currently emerging all over the world. Carbapenemases represent a major public health problem because of the risk of therapeutic impasse and their high epidemic potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom the results of bacteriological examinations reveal the presence of an Enterobacteria strain with reduced susceptibility to carbapenems
* Control : patients ( infected or colonized ) a strain of Enterobacter sensitive to carbapenems immediately isolated after a strain of Enterobacter having decreased susceptibility to carbapenems from the same service and same hospital ( 2 strains susceptible strain with reduced sensitivity).

Exclusion Criteria:

* Duplicate : same strain to a first strain of reduced sensitivity in isolated the same patient during the study period ( same bacterial species , even after characterization resistance mechanism).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing bacteriological samples as part of routine clinical practice during their hospital stay in one of the 6 participating centres. Patients in whom the results of bacteriological examinations reveal the presence of an Enterobacteria strain with reduced susceptibility to carbapenems will be included in this project
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02-02 (Actual); Study Completion 2014-02-02 (Actual)

PRIMARY OUTCOMES:
prevalence of clinical strains of Enterobacteria | 1 year

SECONDARY OUTCOMES:
characterization of the mechanisms responsible for carbapenems resistance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hedi MAMMERI, PhD, Principal Investigator — CHU Amiens
Locations (6):
- France (6):
  - CH Abbeville, Abbeville
  - CHU Amiens, Amiens
  - CH Beauvais, Beauvais
  - CHU Caen, Caen
  - CHU Compiegne, Compiègne
  - CHRU Lille, Lille